CLINICAL TRIAL: NCT02794610
Title: Ocular Penetration of Topical Tacrolimus Eye Drops
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Eye Center and The Eye Foundation for Research in Ophthalmology (Other)
Responsible Party: Principal Investigator, Samir S. Shoughy, MD, FRCS (Glasg.), Principal Investigator, The Eye Center and The Eye Foundation for Research in Ophthalmology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-01(P)
Record Dates: First submitted 2016-05-26; First posted 2016-06-09 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-05

CONDITIONS: Ocular Penetration of Topical Tacrolimus
Keywords: Tacrolimus; Ocular penetration; Topical
MeSH Terms: conditions — Eye Injuries, Penetrating | interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Topical tacrolimus (Experimental): Ten patients will be include. Topical tacrolimus 0.05% will be instilled into the eyes of patients 15 minutes before cataract surgery. Aqueous samples will be collected at the time of cataract surgery and will be subjected to detection of presence and level of tacrolimus.
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — Topical tacrolimus 0.05% eye drops will be instilled into the eyes of patients every minute for 5 minutes. After 15 minutes, at the time of cataract surgery, aqueous samples will be collected and will be subjected to detection of presence and level of tacrolimus.

SUMMARY:
Investigators aim to evaluate the ocular penetration of topical tacrolimus 0.03% eye drops.

Topical tacrolimus 0.03% will be instilled into the eyes of patients 15 minutes before cataract surgery. Aqueous samples will be collected at the time of cataract surgery and will be subjected to detection of presence and level of tacrolimus.

ELIGIBILITY:
Inclusion Criteria:

* Any age or gender
* Patients scheduled for routine cataract surgery
* Clear healthy cornea

Exclusion Criteria:

* Corneal pathology
* Ocular surface disease
* Intraocular inflammation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-05; Primary Completion 2016-06 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Detection of the concentration of tacrolimus ( nanograms/milliliter) in the anterior chamber following ocular topical application. | From date of obtaining the aqueous samples until getting the laboratory results of concentration of topical tacrolimus in the aqueous humor up to 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- The Eye Center, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shoughy SS, Aljassar FM, Tabbara KF. Aqueous penetration of topical tacrolimus. Am J Ophthalmol Case Rep. 2020 Jan 17;17:100582. doi: 10.1016/j.ajoc.2019.100582. eCollection 2020 Mar. PMID 32025589